CLINICAL TRIAL: NCT06169930
Title: Development and Validation of A Overall Survival Prediction Model for Esophageal Squamous Cell Carcinoma: A Novel pN Classification
Brief Title: Development and Validation of a Survival Prediction Model for Esophageal Cancer Patients After Esophagectomy
Acronym: OSmodel
Status: Completed | Type: Observational
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, MD, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCH-TS2207
Record Dates: First submitted 2023-12-03; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Survivorship
Keywords: survival; esophgeal cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk
  Interventions: Other: This was an observational study without any intervention
- low-risk
  Interventions: Other: This was an observational study without any intervention

INTERVENTIONS:
Other: This was an observational study without any intervention — This was an observational study without any intervention

SUMMARY:
In this retrospective study, we analyzed data from the Sichuan Cancer Hospital & Institute Esophageal Cancer Case Management Database (SCH-ECCM Database) from January 2010 to December 2017. Our study focused on examining the clinicopathological characteristics, lymph node removal at each station, and treatment details of patients with esophageal squamous cell carcinoma (ESCC) who underwent esophagectomy. Using this data, we developed a prediction model for OS by considering a combination of clinical characteristics and details of lymphadenectomy variables.

DETAILED DESCRIPTION:
In this retrospective study, we analyzed data from the Sichuan Cancer Hospital & Institute Esophageal Cancer Case Management Database (SCH-ECCM Database) from January 2010 to December 2017. Our study focused on examining the clinicopathological characteristics, lymph node removal at each station, and treatment details of patients with esophageal squamous cell carcinoma (ESCC) who underwent esophagectomy. Using this data, we developed a prediction model for OS by considering a combination of clinical characteristics and details of lymphadenectomy variables. Additionally, the receiver operating characteristic curve demonstrated an area under the curve greater than 0.7 at 1, 3, and 5 years in both the verification and training groups. Furthermore, Kaplan-Meier (K-M) curves showed that our model effectively distinguished between high- and low-risk groups (p < 0.01).

ELIGIBILITY:
Inclusion criteria:

* Patients underwent esophagectomy at our hospital.

Exclusion criteria:

* pathology confirmed a non-squamous cell carcinoma,
* the tumor was located outside of the thoracic region,
* R1/R2 resection was performed indicating incomplete tumor removal,
* evidence of distant tumor metastasis was observed, or
* they underwent preoperative neoadjuvant therapy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the Sichuan Cancer Hospital & Institute Esophageal Cancer Case Management Database (SCH-ECCM Database) from January 2010 to December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 2957 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Survival | April 2022-April 2024
  Overall survival (OS) was defined as the time from the month and year of surgery until death or the last follow-up in April 2022.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No